CLINICAL TRIAL: NCT01816529
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of Diltiazem Hydrochloride 2% Cream in Healthy Subjects Using a Repeat Insult Patch Test Design
Brief Title: Topical Safety Study of Topical Diltiazem Hydrochloride
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VEN307-DERM-001
Record Dates: First submitted 2013-03-18; First posted 2013-03-22 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-07

CONDITIONS: Diltiazem Skin Sensitivity.
MeSH Terms: interventions — Diltiazem; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Topical Diltiazem Hydrochloride 2% Cream (Experimental): 0.2 g cream applied topically to the infrascapular area of the back under occlusive patch conditions, 3 times weekly for 3 weeks and one time at Challenge. A total of 10 patch applications over 6-8 weeks.
  Interventions: Drug: Diltiazem Hydrochloride 2% Cream
- Vehicle Cream (Placebo Comparator): 0.2 g cream applied topically to the infrascapular area of the back under occlusive patch conditions, 3 times weekly for 3 weeks and one time at Challenge. A total of 10 patch applications over 6-8 weeks.
  Interventions: Drug: Vehicle Cream
- 0.1% solution of sodium lauryl sulfate (SLS) (Active Comparator): 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions, 3 times weekly for 3 weeks and one time at Challenge. A total of 10 patch applications over 6-8 weeks.
  Interventions: Drug: 0.1% solution of sodium lauryl sulfate (SLS)
- 0.9% Saline (Placebo Comparator): 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions, 3 times weekly for 3 weeks and one time at Challenge. A total of 10 patch applications over 6-8 weeks.
  Interventions: Drug: Saline (0.9%)

INTERVENTIONS:
Drug: Diltiazem Hydrochloride 2% Cream — 0.2 g applied topically to the infrascapular area of the back.
  Arms: Topical Diltiazem Hydrochloride 2% Cream
Drug: Vehicle Cream — Vehicle Cream, 0.2 g (contains no active pharmaceutical ingredient) applied topically to the infrascapular area of the back.
  Arms: Vehicle Cream
Drug: 0.1% solution of sodium lauryl sulfate (SLS) — 0.2 mL applied topically to the infrascapular area of the back will serve as a positive control.
  Arms: 0.1% solution of sodium lauryl sulfate (SLS)
Drug: Saline (0.9%) — 0.2 mL applied topically to the infrascapular area of the back will serve as a negative control.
  Arms: 0.9% Saline

SUMMARY:
The goal of this study will be to determine the potential of Diltiazem Hydrochloride 2% Cream to induce sensitization by repeated topical application to the skin of healthy subjects under controlled conditions.

DETAILED DESCRIPTION:
The primary objective of this study will be to determine the potential of Diltiazem Hydrochloride 2% Cream and its vehicle to induce sensitization by repeated topical application to the skin of healthy subjects under controlled conditions. In addition, the irritation potential of the investigational products will be assessed during the Induction Phase and safety will be assessed by evaluation of any adverse events (AEs) reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females (to be confirmed by medical history);
* Are 18 years of age or older;
* In the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
* In the case of females of childbearing potential: have a negative urine pregnancy test (UPT) at Screening, and are willing to submit to a pregnancy test at the end of study (EOS);
* Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
* Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema;
* Read, understand, and provide signed informed consent.

Exclusion Criteria:

* Have sick sinus syndrome except in the presence of a functioning ventricular pacemaker (confirmed via medical history);
* Have second-or third-degree AV block except in the presence of a functioning ventricular pacemaker (confirmed via medical history);
* Have hypotension (less than 90 mm Hg systolic, determined by performing vital signs);
* Have acute myocardial infarction and pulmonary congestion documented by x-ray (confirmed via medical history);
* Have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction;
* Are not willing to refrain from using topical/systemic analgesics such as aspirin (daily use of 81 mg aspirin is acceptable), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
* Are using systemic/topical corticosteroids for 3 weeks prior to and during the study, or systemic/topical antihistamines for 72 hours prior to and during the study;
* Are using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications;
* Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions, or similar products on the back during the study;
* Have psoriasis and/or active atopic dermatitis/eczema;
* Are females who are pregnant, plan to become pregnant during the study, or are breast-feeding a child;
* Have a known sensitivity to constituents present in the material being evaluated;
* Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* Have received treatment for any type of internal cancer within 5 years prior to study entry;
* Have a history of, or are currently being treated for skin cancer;
* Are currently participating in any clinical testing,
* Have any known sensitivity to adhesives; and/or
* Have received any investigational treatment(s) within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Determine the potential of Diltiazem Hydrochloride 2% Cream to induce sensitization by repeated topical application to the skin of healthy subjects under controlled conditions. | 6 weeks after the first topical application
  A total cumulative irritation score for each subject and product will be calculated by summing each individual's scores on each of the 9 evaluation days in the Induction Phase. Cumulative irritancy during Induction will be quantified by means of the cumulative irritancy index (CII), defined as the mean of irritation scores received during the Induction Phase (9 readings). The determination of dermal sensitization potential will be based on specific scoring criteria derived from observations in the Challenge Phase of the study and confirmed in the Rechallenge Phase, if necessary. The recurrence of a cutaneous response at Rechallenge equivalent to or more severe than that observed at challenge will be considered indicative of a sensitization reaction. The observation of such a response in even a single subject suggests that the test product may have the potential to cause hypersensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Paramus, New Jersey, United States